CLINICAL TRIAL: NCT05348707
Title: Impact of Covid-19 Pandemic on the Epidemiology of Rhinovirus
Brief Title: Impact of Covid-19 on Rhinovirus Epidemic
Acronym: IPCoRV
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 502_2
Record Dates: First submitted 2022-02-17; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-02

CONDITIONS: Rhinovirus
Keywords: Rhinovirus epidemic; SARS-CoV2/Rhinovirus interaction; Children; Non-pharmacological-interventions; Bronchiolitis; Asthma; Pneumonia; Fever; Meningitis; Rhinovirus infection in children less than 1 years of age
MeSH Terms: conditions — Bronchiolitis; Asthma; Pneumonia; Fever; Meningitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pre Covid 19 cohort: Infants hospitalized in the Pediatric Department of the " Hôpital Femme Mère Enfant ", Lyon, France with a RT-PCR positive for Rhinovirus from 17th March 2019 to 16th March 2020.
  Interventions: Other: epidemiology
- Per Covid 19 cohort year 1: Infant hospitalized in the Pediatric Department of the " Hôpital Femme Mère Enfant ", Lyon, France with a RT-PCR positive for Rhinovirus from 17th March 2020 to 16th March 2021. The need to recruit patients for an additional per-covid year (from 17th March 2021 to 16th March 2022) will be evaluated after the data from the first 2 years of recruitment are available.
  Interventions: Other: epidemiology
- Per Covid 19 cohort, year 2: Infants hospitalized in the Pediatric Department of the " Hôpital Femme Mère Enfant ", Lyon, France with a RT-PCR positive for Rhinovirus from 17th March 2021 to 16th March 2022. The need to recruit patients for this additional cohort will be evaluated after the data from the first 2 years of recruitment are available and analyzed.
  Interventions: Other: epidemiology

INTERVENTIONS:
Other: epidemiology — To review medical records to describe diagnosis and severity of the disease.
  Other Names: Medical record analysis
Other: epidemiology — To compare pre and per Covid-19 epidemics in terms of numbers of admissions and proportion of severe disease.
  Other Names: Comparison of cohorts

SUMMARY:
Rhinovirus (RV) has long been known as the main etiological agent of "common colds" among children and adults. Indeed, RV is involved in more than 50% of upper respiratory tract infections (URTIs), mostly characterized by nasal congestion, rhinorrhea, sore throat and cough. RV can also cause mild to severe lower respiratory tract infections (LRTIs) such as acute bronchiolitis, pneumonia and exacerbations of underlying chronic lung diseases. RV circulates worldwide, especially in temperate climate zones (i.e. many areas of the USA and Europe) and is responsible for annual outbreaks from early fall to the end of spring.

The covid-19 pandemic in 2020 seemed to interfere with the usual seasonal epidemics. For example, the winter Respiratory Syncytial Virus (RSV) epidemic in Lyon, France, was delayed for several months and reduced by half in terms of incidence of hospitalization cases. This can be explained by the widespread deployment of barrier gestures and social distancing measures, known as "non pharmacological interventions" (NPI).

However, the Covid-19 pandemic doesn't seem to have the same reducing impact on Rhinovirus epidemic. A better understanding of viral interactions and factors influencing RV epidemiology as well as the identification of populations at greater risk are required to improve preventive strategies and reduce the burden of Rhinovirus.

ELIGIBILITY:
Inclusion Criteria:

* - Child hospitalized at the " Hopital Femme Mere Enfant ", Lyon, France
* Positive rhinovirus-PCR

Exclusion Criteria:

* - parent's refusal to participate

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Child hospitalized at the " Hopital Femme Mere Enfant ", Lyon, France
  - Positive rhinovirus-PCR
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Evolution of the number of children hospitalized for a Rhinovirus-infection in the period of pre Covid-19 pandemic. | From one year before the SARS-CoV-2 pandemic until the beginning of the SARS-CoV-2 pandemic
  Description of number of clinical picture cases for pre-SARS-CoV-2 pandemic year.
Evolution of the number of children hospitalized for a Rhinovirus-infection in the period of per-Covid-19 pandemic. | From the beginning of the SARS-CoV-2 pandemic until one year latter
  Description of number of clinical picture cases for per-SARS-CoV-2 pandemic year.

IPD SHARING:
Plan to Share IPD: Undecided